CLINICAL TRIAL: NCT07097870
Title: Study of Clinical and Laboratory Predictors of Hepatocellular Carcinoma in Post-HCV Cirrhotic Patients After Sustained Virologic Response.
Brief Title: Predictors of HCC in Post-HCV Cirrhotic Patients After SVR
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zakaria Saeed Gerges Awad, Internal Medicine Resident Doctor, Sohag University
Other Study IDs: Soh-Med--25-7-12MS
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: HCV; Sustained virologic response; HCC; SVR; liver cirrhosis; DAA; Direct acting antivirals
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: SVR patients who developed HCC
- Controls: SVR patients who did not develop HCC

SUMMARY:
This study aims to identify clinical and laboratory factors that predict the occurrence of hepatocellular carcinoma (HCC) in Egyptian cirrhotic patients after achieving a sustained virologic response (SVR) to hepatitis C virus (HCV) treatment. This is a retrospective, two-center, case-control study that will include 132 cases and 264 controls. Variables to be analyzed include demographics, liver disease status, metabolic comorbidities, lifestyle factors, medications, as well as laboratory parameters and non-invasive scoring systems.

DETAILED DESCRIPTION:
Introduction:

Hepatocellular carcinoma (HCC) is a highly fatal cancer with a global 5-year survival rate of less than 20%. In Egypt, HCC is the most common cancer in men and the leading cause of cancer-related death, primarily due to the historically high prevalence of Hepatitis C Virus (HCV). While sustained virologic response (SVR) after direct-acting antiviral (DAA) therapy significantly reduces the risk of HCC, it can still occur, especially in patients with advanced fibrosis or cirrhosis. This necessitates continued HCC surveillance post-HCV cure.

Aim of Work:

To study various clinical and laboratory predictors of hepatocellular carcinoma in Egyptian cirrhotic patients after achieving sustained virologic response.

Methodology:

Study Design: Retrospective, two-center case-control study.

Setting & Period: Two tertiary hepatology centers: Sohag University Hospital and Sohag Oncology Center.

SVR was achieved between January 1, 2016 - December 31, 2019

Participants:

Cases: SVR patients who developed HCC

Inclusion Criteria: (1) age ≥ 18 y; (2) HCV related cirrhosis; (3) SVR12 after DAA; (4) radiologic or histologic HCC diagnosis ≤30 Jun 2025

Exclusion Criteria: (1) non HCV cirrhosis or combined HCV-HBV cirrhosis; (2) HCC <6 months before SVR; (3) concomitant cholangiocarcinoma

Controls: SVR patients who did not develop HCC Inclusion Criteria: As above plus,

≥36 months post SVR without HCC

Exclusion Criteria: Same as cases, plus loss to follow-up before 36 months

Sample Size: Using Fleiss' formula yields 120 cases & 240 controls (360 total). Adding 10 % for incomplete charts ⇒ 132 cases & 264 controls (≈ 400 subjects).

Variables to Study:

Clinical Predictors: Demographics (Age, Sex, Residence), Liver disease status (History of decompensation, Splenomegaly, Time since SVR), Metabolic comorbidities (Diabetes mellitus, Obesity/BMI, Dyslipidemia, HTN), Lifestyle factors (Smoking, Alcohol use), Medications (Statins, Metformin, Aspirin).

Laboratory Predictors: Platelet count, AST, ALT, AST/ALT ratio, Albumin, Total bilirubin, INR, Alpha-fetoprotein (AFP), HbA1c, Creatinine, Urea, GGT, and ALP.

Non-Invasive Scoring Systems: Child-Pugh Score, MELD Score, FIB-4 Score, ALBI Score, APRI, AAR (AST/ALT ratio).

Ethical Considerations: Approved by IRBs of both centers. Waiver of informed consent granted (retrospective chart review, minimal risk).

Duration: 6 months

ELIGIBILITY:
Inclusion Criteria:

* for cases:

  1. age ≥ 18 y;
  2. HCV related cirrhosis;
  3. SVR12 after DAA;
  4. radiologic or histologic HCC diagnosis ≤30 Jun 2025
* for controls: As above plus, ≥36 months post SVR without HCC

Exclusion Criteria:

* for cases:

  1. non HCV cirrhosis or combined HCV-HBV cirrhosis;
  2. HCC <6 months before SVR;
  3. concomitant cholangiocarcinoma
* for controls: Same as cases, plus, loss to follow up before 36 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-HCV cirrhotic patient from Egypt, after achieving SVR 12 (between 2016-2019) who did (cases) or did not (controls) develop HCC
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
occurrence of hepatocellular carcinoma (HCC) | from SVR12 achievement to 6-9 years later (time of data collection)
  measure occurrence of HCC in post-HCV liver cirrhosis after achieving SVR, by comparing cases to controls

CONTACTS AND LOCATIONS:
Overall Officials: Usama A Arafa, PhD, Study Chair — Faculty of Medicine, Sohag university; Ali M Hussein, PhD, Study Director — Faculty of Medicine, Sohag university
Locations (1):
- Faculty of Medicine, Sohag Univesity, Sohag, Egypt